CLINICAL TRIAL: NCT04563572
Title: Determine AF Burden With PPG Trial - Detection and Quantification of Episodes of Atrial Fibrillation Using a Cloud Analytics Service Connected to a Wearable With Photoplethysmographic (PPG) Sensor
Brief Title: Determine AF Burden With PPG Trial - Detection and Quantification of Episodes of Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Preventicus GmbH (Industry); Manufacture Modules Technologies SA (Unknown); GETEMED GmbH (Unknown); Eurostars (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-01983
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Wearables; AF Burden; Photoplethysmography (PPG); Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Participants will receive a PPG sensor in form of a smartwatch or a bracelet and will be instructed to wear them continuously for 48 hours. Assigning patients to the smartwatch or the bracelet group will occur in an alternating fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPG Smartwatch (Experimental): The Preventicus Heartbeats algorithm ist a certified tool for detection of Atrial Fibrillation. It differentiates accurately between regular rhythm, single premature beats and the absolute arrhythmia concordant with AF. The Preventicus algorithm is device-agnostic, meaning that any wearable device capable of recording PPG-signals can be used for data collection.
  CardioWatch 287 is a novel non-invasive monitoring device manufactured by the MMT company. The device monitors heart rhythm, heart rate (HR) and respiratory rate (RR) based on peripheral PPG signal.
  In this arm, we will test the quality of the algorithm integrated into the smartwatch.
  Interventions: Device: PPG Smartwatch
- PPG Bracelet (Experimental): The Preventicus Heartbeats algorithm ist a certified tool for detection of Atrial Fibrillation. It differentiates accurately between regular rhythm, single premature beats and the absolute arrhythmia concordant with AF. The Preventicus algorithm is device-agnostic, meaning that any wearable device capable of recording PPG-signals can be used for data collection.
  A PPG-sensor is also integrated into a bracelet "Basler Band" manufactured by the MMT company, which is a simplified multisensory device.
  In this arm, we will test the quality of the algorithm integrated into the bracelet.
  Interventions: Device: PPG Smartwatch

INTERVENTIONS:
Device: PPG Smartwatch — Participants will then receive a PPG sensor in form of a smartwatch) model and will be instructed to wear them continuously for 48 hours. Simultaneously, a 48-hour Holter ECG will be performed. Start time on the PPG-sensor and the Holter ECG will be matched and continuous heart rhythm and -rate monitoring will be initiated. Patients will wear the devices over a 48-hour period of time.

SUMMARY:
In this prospective single-center trial, a wearable photoplethysmographic (PPG) sensor coupled with a cloud analytics service will be used to detect and quantify atrial fibrillation (AF) episodes in patients with known paroxysmal AF. Patients will simultaneously receive the PPG sensor in form of a smartwatch or bracelet and a Holter ECG for 48 hours. Correctly identified AF episodes and AF burden determined by both methods will be compared.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac arrhythmia and a major risk factor for cerebrovascular insults. Paroxysmal AF is defined as an episode of AF that terminates spontaneously or with intervention within 7 days. Patients with AF may present with palpitations, shortness of breath or sensation of light-headedness but asymptomatic episodes are also possible, especially in paroxysmal AF. The lack of continuous heart rate monitoring options makes early diagnosis of paroxysmal AF challenging. In this prospective single-center trial, the PPG wearable Corsano CardioWatch 287 sensor will be used to conduct continuous heart rate and -rhythm monitoring in patients with known paroxysmal AF. Collected data will then be analysed using a Cloud Analytics Service (Preventicus Heartbeats algorithm) and compared with data from simultaneously obtained 48-hour Holter ECG. Correctly identified AF episodes, their cumulative duration per 48 hours (AF burden) and the number of asymptomatic episodes will be assessed. In the primary analyses, the sensitivity of the PPG analysing algorithm to detect AF episodes is estimated by performing a logistic regression on detection (yes/no) with only an intercept as predictor, which is then translated to a proportion (the sensitivity). In the secondary analyses we are comparing the cumulative duration of AF episodes over 48 hours (AF burden) obtained with the PPG-sensor and Holter-ECG. In summary, the purpose of the study is to evaluate the performance and efficacy of the wearable PPG sensor and the cloud analytics service in detecting and quantifying AF episodes in patients with known history of paroxysmal AF.

ELIGIBILITY:
Inclusion Criteria:

* Known paroxysmal atrial fibrillation
* Patient ≥ 18 years old
* Written informed consent as documented by signature from the patient

Exclusion Criteria:

* Cardiac implanted electronic device (Pacemaker, ICD)
* Smartwatch/Bracelet and/or ECG device cannot be worn due to comprehensible reasons (allergic reactions, wounds, amputations, other)
* Patients unable or not willing to sign informed consent Significant mental or cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Number of AF episodes | 48 hours
  Number of detected atrial fibrillation episodes by the PPG sensor and Preventicus Heartbeats algorithm during the 48h trial period compared to the Holter ECG.

SECONDARY OUTCOMES:
AF Burden | 48 hours
  Cumulative duration of AF episodes
Asymptomatic AF episodes | 48 hours
  Number of asymptomatic AF episodes

CONTACTS AND LOCATIONS:
Overall Officials: Jens Eckstein, MD, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Universitiy Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reissenberger P, Serfozo P, Piper D, Juchler N, Glanzmann S, Gram J, Hensler K, Tonidandel H, Borlin E, D'Souza M, Badertscher P, Eckstein J. Determine atrial fibrillation burden with a photoplethysmographic mobile sensor: the atrial fibrillation burden trial: detection and quantification of episodes of atrial fibrillation using a cloud analytics service connected to a wearable with photoplethysmographic sensor. Eur Heart J Digit Health. 2023 Jul 6;4(5):402-410. doi: 10.1093/ehjdh/ztad039. eCollection 2023 Oct. PMID 37794868